CLINICAL TRIAL: NCT03674359
Title: Performance of the Dosage of Plasma 1, 3-β-D-glucan (BDG) for the Diagnosis of Candidemia in Intensive Care Patients: A Prospective, Multicenter Study
Brief Title: Dosage of Plasma 1, 3-β-D-glucan for the Diagnosis of Candidemia.
Acronym: BDG-REA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P170926J
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-12

CONDITIONS: Infection, Fungal
Keywords: 1, 3-β-D-glucan, Candidemia, Intensive Care Unit
MeSH Terms: conditions — Mycoses; Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, plasma for dosage of 1, 3-β-D-glucan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients hospitalized in intensive care, meeting the inclusion criteria. BDG analysis
  Interventions: Diagnostic Test: BDG analysis

INTERVENTIONS:
Diagnostic Test: BDG analysis — BDG analysis

SUMMARY:
Systematic and repeated dosing (3 times weekly) of 1,3-β-D-glucan (BDG), associated with blood cultures and fungal mapping (twice a week) for the patients hospitalized in intensive care. The diagnosis of candidemia is defined as the 1st positive blood culture for Candida spp.

The dosage of BDG will be considered positive if the value is at least or equal to 80 pg/ml.

DETAILED DESCRIPTION:
The candidemia is the 3rd cause of sepsis in intensive care unit and a serious problem because the high mortality remains (> 50%) despite the new treatments by echinocandins.

A single positive blood culture is sufficient for diagnosis, but the sensitivity of blood cultures is only 50 to 70 percent. Clinical signs are unspecific and do not guide the diagnosis. If treatment started early, 12 hours after the 1st positive blood culture collection the mortality is 10%. Recently, the incidence of candidemia in intensive care unit has increased in France as in other countries as. From these different elements (frequency, mortality, early diagnosis, little specific clinical signs), it is easy to understand the approach that has prevailed for many years, which is to define the profile of the patients at risk of candidemia in intensive care unit. Currently, there are several predictive factors of occurrence of a candidemia in intensive care unit. They are represented by the index of colonization, very high risk factors (FTHR) and Candida score (CS).

Predictive factors of occurrence of candidemia have led to the concept of preemptive or empirical treatment, the aim is to being avoid the occurrence of candidemia.

However, the ability of these factors to predict the occurrence of a candidemia is not satisfactory, explaining in part the mortality rate.

In the light of current knowledge, including the predictive factors of occurrence of candidemia in intensive care patients, a better selection of patients likely to develop candidemia remains to this day, a crucial issue. Several teams have been interested in the evaluation of various bio-markers, including the (1,3) - β - D-glucan (BDG), to optimize decision-making in intensive care patients at risk of candidemia in front of:

* the increased frequency of candidemia,
* poorly discriminating predictive factors,
* no specific clinical signs,
* the low sensitivity of blood culture,
* and the impact of early treatment.

To clarify the role of BDG as a predictive factor of candidemia, all patients hospitalized in intensive care unit, meeting the criteria for inclusion and exclusion, will be followed, from day 4 of hospitalization or from the beginning of antifungal treatment between the admission in intensive care unit and day 4, until the exit of intensive care unit or until day30 of hospitalization in intensive care unit.

The dosage of BDG and blood cultures will be performed on day 4 of hospitalization or before the beginning of antifungal treatment between the admission in intensive care unit and the 4th day, then 3 times a week, until day 30.

A before the beginning of antifungal treatment between the admission to intensive care unit and the 4th day of hospitalization, then twice a week, maximum until day30.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients Under mechanical ventilation (MV), antibiotic (AB) And with a central venous catheter (CVK)
* inclusion at day 4 of hospitalization or from establishing of antifungal treatment between admission to the Intensive Care Unit (ICU) and day 4
* Affiliation to the social security system.
* Signed informed consent

Exclusion Criteria:

* Antifungal therapy at the admission in intensive care unit
* Patient whose inclusion life expectancy is less than 72 h
* Patient being treated for Pneumocystis carinii pneumonia (PCP)
* Pregnant or breastfeeding woman
* Neutropenia: < 500 nuclear neutrophil / mm3
* Patients under ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18, hospitalized in intensive care unit, under mechanical ventilation, antibiotics and with a central venous catheter, excluding pregnant or breastfeeding women.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Determine the sensitivity and specificity of the BDG for the diagnosis of candidemia in intensive care unit patients. | 30 day after inclusion
  Systematic and repeated dosing , for the diagnosis of candidemia (1st positive blood culture for Candida spp).
  Dosage of BDG will be considered positive if a dosage is at least equal to 80 pg/ml or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe KAROUBI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hopital Avicenne, Bobigny
  - Hôpital Louis Mourier, Colombes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lortholary O, Renaudat C, Sitbon K, Madec Y, Denoeud-Ndam L, Wolff M, Fontanet A, Bretagne S, Dromer F; French Mycosis Study Group. Worrisome trends in incidence and mortality of candidemia in intensive care units (Paris area, 2002-2010). Intensive Care Med. 2014 Sep;40(9):1303-12. doi: 10.1007/s00134-014-3408-3. Epub 2014 Aug 6. PMID 25097069
- [Result] Clancy CJ, Nguyen MH. Finding the "missing 50%" of invasive candidiasis: how nonculture diagnostics will improve understanding of disease spectrum and transform patient care. Clin Infect Dis. 2013 May;56(9):1284-92. doi: 10.1093/cid/cit006. Epub 2013 Jan 11. PMID 23315320
- [Result] Morrell M, Fraser VJ, Kollef MH. Delaying the empiric treatment of candida bloodstream infection until positive blood culture results are obtained: a potential risk factor for hospital mortality. Antimicrob Agents Chemother. 2005 Sep;49(9):3640-5. doi: 10.1128/AAC.49.9.3640-3645.2005. PMID 16127033
- [Result] Posteraro B, De Pascale G, Tumbarello M, Torelli R, Pennisi MA, Bello G, Maviglia R, Fadda G, Sanguinetti M, Antonelli M. Early diagnosis of candidemia in intensive care unit patients with sepsis: a prospective comparison of (1-->3)-beta-D-glucan assay, Candida score, and colonization index. Crit Care. 2011;15(5):R249. doi: 10.1186/cc10507. Epub 2011 Oct 22. PMID 22018278